CLINICAL TRIAL: NCT04565431
Title: Biomarker for Cognitive Fatigue Using Functional Imaging in Multiple Sclerosis
Brief Title: Examining Effects of Tysabri on Cognitive Fatigue Using fMRI
Status: Recruiting | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: St. Barnabas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: US-TYS-11640
Record Dates: First submitted 2020-08-25; First posted 2020-09-25 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Cognitive Fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group 1: Multiple Sclerosis: Individuals with RRMS who are going to be starting Tysabri as determined by Neurologist as part of clinical care.
  Intervention: Drug: Tysabri
  Interventions: Drug: Tysabri
- Group 2: Healthy Controls: Healthy individuals who are age, gender and education matched to the MS group.

INTERVENTIONS:
Drug: Tysabri — Participants with RRMS who are planning to begin treatment with Tysabri will be compared to a group of healthy individuals who are matched for age, gender, and education.
  Groups: Group 1: Multiple Sclerosis

SUMMARY:
The purpose of this research study is to investigate the effectiveness of Tysabri on cognitive fatigue in persons with Relapsing-Remitting Multiple Sclerosis (RRMS). Cognitive fatigue is the kind of fatigue that occurs after intense mental concentration as after a session of problem solving.

DETAILED DESCRIPTION:
The researchers aim is to investigate the effects of Tysabri on cognitive fatigue and on specific brain areas that have been shown to underlie cognitive fatigue in individuals with RRMS. The researchers will investigate the effects on the cognitive fatigue that develops during the performance of a demanding task and also on how cognitive fatigue changes as a function of duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64
* Diagnosed with Relapsing-Remitting Multiple Sclerosis or a healthy volunteer
* If diagnosed with MS: has been newly prescribed Tysabri, but has not yet started taking the medication
* Can read and speak English fluently

Exclusion Criteria:

* History of head injury, stroke, seizures, or any other significant neurological event other than MS
* Flare up of MS symptoms within the past month
* History of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder
* Pacemaker or other implanted electrical device, brain stimulator, aneurysm clip (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments
* Left-handed.
* Not able to have an MRI

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals diagnosed with Relapsing-Remitting Multiple Sclerosis and Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brain activation (BOLD signal) | Measured by change between 2 time points (baseline and six months after intervention)
  A change in brain activation as measured with functional magnetic resonance imaging through blood oxygen level dependent signal will be measured in association with cognitive fatigue (as measured by the Visual Analogue scale during performance of the modified Symbol Digit Modality Task and Modified Fatigue Impact Scale).

SECONDARY OUTCOMES:
Fatigue onset (SDMT) | Measured by change between 2 time points (baseline and six months after intervention)
  A change in the speed with which modified Symbol Digit Modality Task (a cognitively demanding task) induces fatigue in MS (as measured by the Visual Analogue scale)
Fatigue onset | Measured by change between 2 time points (baseline and six months after intervention)
  A change in brain activation as measured with functional magnetic resonance imaging through blood oxygen level dependent signal will be measured in association with cognitive fatigue (as measured by the Modified Fatigue Impact Scale)

CONTACTS AND LOCATIONS:
Overall Officials: John DeLuca, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States